CLINICAL TRIAL: NCT02082964
Title: The Effect of SCIM on Neonatal Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, fatemeh erfanian, instructor of midwifery Ph.D student, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: training
Record Dates: First submitted 2014-02-13; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Pregnancy
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SCIM (Experimental): after lecture students had rotation in 6 groups through 6 stations, trained and practiced under supervision of 6 instructors about Initial Steps, Positive Pressure Ventilation(PPV), Intubation, Chest Compressions, Medications and management of advanced resuscitation
  Interventions: Other: SCIM
- video (Experimental): video about neonatal resuscitation presented then students repeated the video. Workshops was based on NRP and lasted 6 hours for each group the contentof the video was based on the educational content of the course.
  Interventions: Other: video

INTERVENTIONS:
Other: SCIM — after lecture students had rotation in 6 groups through 6 stations, trained and practiced under supervision of 6 instructors about Initial Steps, Positive Pressure Ventilation(PPV), Intubation, Chest Compressions, Medications and management of advanced resuscitation
  Arms: SCIM
Other: video — video about neonatal resuscitation presented then students repeated the video. Workshops was based on NRP and lasted 6 hours for each group the contentof the video was based on the educational content of the course
  Arms: video

SUMMARY:
In this randomized controlled trial 48 students were randomly allocated in three groups SCIM, Video training (VT) and control group(no training). They had a workshops based on NRP and lasted 6 hours for each group. Before and after the workshops and one month later all students participated in a 7 station OSCE..

ELIGIBILITY:
Inclusion Criteria:

healthy, without any history of severe stress in the past 6 months prior to the study. Accepts Healthy Volunteers

Exclusion Criteria:severe stress

-

Ages: 22 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
education | 3 months
  after educational course for each group (SCIM and Video), students' competency in neonatal resuscitation would be evaluated through an OSCE in each group. the competency between group (before and after education) and in each group would be comapared before and after education.

CONTACTS AND LOCATIONS:
Locations (1):
- Mashhad, Iran